CLINICAL TRIAL: NCT02057367
Title: The Effect of Pre-incisional Anterior Scalp Block on Intraoperative Opioid Consumption in Adult Patients Undergoing Elective Craniotomy to Remove Tumor: A Prospective Randomized Controlled
Brief Title: Scalp Nerve Block and Opioid Consumption in Brain Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Department of Anesthesiology, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANE2556-01510
Record Dates: First submitted 2013-09-26; First posted 2014-02-07 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Brain Tumour
Keywords: supratentorial brain tumour; craniotomy
MeSH Terms: conditions — Brain Neoplasms | interventions — Saline Solution; PAVE protocol 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scalp block with 0.5% plain marcaine (Experimental): Anterior scalp block with 0.5% plain Marcaine 20 ml.
  Interventions: Drug: Scalp block with 0.5% plain Marcaine
- Scalp block with 0.9% normal saline (Placebo Comparator): Anterior scalp block with 0.9% normal saline 20 ml.
  Interventions: Drug: Scalp block with 0.9% normal saline

INTERVENTIONS:
Drug: Scalp block with 0.5% plain Marcaine — Anterior scalp block will be done by using 0.5% plain Marcaine 20 ml.
  Other Names: Code 1
  Arms: Scalp block with 0.5% plain marcaine
Drug: Scalp block with 0.9% normal saline — Anterior scalp block will be done by using 0.9% normal saline 20 ml.
  Other Names: Code 2
  Arms: Scalp block with 0.9% normal saline

SUMMARY:
Anterior scalp block with 0.5% plain Marcaine 20 ml. may reduce the intraoperative opioid consumption in neurosurgical patients who undergoing the supratentorial craniotomy compared to those who receive 0.9% normal saline solution (placebo).

DETAILED DESCRIPTION:
Anterior scalp block with 0.5% plain Marcaine 20 ml. may reduce the intraoperative opioid consumption in neurosurgical patients who undergoing the supratentorial craniotomy compared to those who receive 0.9% normal saline solution (placebo).

A Prospective Randomized Double Blind Control

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have supratentorial brain tumor
2. Patients have been scheduled to undergo an elective craniotomy to remove tumor in any surgical position
3. Patients have been general anesthetized with endotracheal intubation and control ventilation
4. Patients who have provided consent for the participation in the research and for the use of their medical record in research

Exclusion Criteria:

1. Pregnant patients
2. Patients who have a history of local anesthetic allergy and/ or anaphylaxis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Intraoperative opioid consumption | During the supratentorial craniotomy surgery
  The overall intravenous fentanyl consumption (microgram/ kilogram) during the surgery. The decision to administer fentanyl is guided by the changes of blood pressure and/ or heart rate greater than 20% from baseline level.

SECONDARY OUTCOMES:
systolic blood pressure change | within 5 minutes after skull pin insertion
  The maximal systolic blood pressure within the first 5 minutes after skull pin insertion will be recorded.
  The systolic blood pressure change from baseline will be calculated. The unit is mmHg.
Heart rate change | within 5 minutes after skull pin insertion
  The maximal heart rate within the first 5 minutes after skull pin insertion will be recorded.
  The heart rate change from baseline level will be calculated. The unit is beats per minute.

OTHER OUTCOMES:
extubation | end of surgery, before transferring to the intensive care unit
  The rate of immediate extubation before transferring to the intensive care unit (ICU) compared between patients who received 0.5% plain Marcaine and 0.9% normal saline solution.

CONTACTS AND LOCATIONS:
Overall Officials: Pathomporn Pin-on, M.D., Principal Investigator — Chiang Mai University
Locations (1):
- Chiang Mai University, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No